CLINICAL TRIAL: NCT04213482
Title: Evaluating Radiomorphometric Indices and Fractal Dimension of the Pediatric Oncology Patients on Panoramic Images
Status: Completed | Type: Observational
Sponsor: Nuh Naci Yazgan University (Other)
Responsible Party: Principal Investigator, Hatice Cansu Kış, Assistant Professor, Nuh Naci Yazgan University
Other Study IDs: 2018/209
Record Dates: First submitted 2019-12-23; First posted 2019-12-30 (Actual); Last update posted 2019-12-30 (Actual); Status verified 2019-12

CONDITIONS: Oncology; Bone Loss
Keywords: pediatric oncology; fractal analysis; panoramic mandibular indices; radiotherapy; chemotherapy
MeSH Terms: conditions — Neoplasms; Bone Diseases, Metabolic | interventions — Radiography, Panoramic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- oncology patients: For this study, panoramic images were taken from pediatric patients who received radiotherapy and/or chemotherapy because of any oncologic disease.
  Interventions: Radiation: Panoramic Radiography
- healthy: panoramic images of patients(pediatric) who have no systemic disease were collected from the archive of dental radiology clinic of the university hospital.
  Interventions: Radiation: Panoramic Radiography

INTERVENTIONS:
Radiation: Panoramic Radiography — Diagnostic Panoramic Dental Radiographs were taken.

SUMMARY:
This study evaluated pediatric oncology patients in terms of quality of bone and determine any relation between bone quality and radiotherapy/chemotherapy. The alternative hypothesis is that the bone quality of the oncology patients who received radiotherapy/chemotherapy is lower than the control group.

DETAILED DESCRIPTION:
Cancer is the abnormal and uncontrolled proliferation of certain tissues in the body for a reason that cannot be determined yet. Childhood cancers occur between 0-17 years of age, and follow-up and treatment of these patients are performed in pediatric oncology services. Diagnosis in childhood cancers can be made by clinical examination as well as blood tests and examination of tissue samples. There are also some imaging methods used for diagnosis; ultrasonography, computed tomography, magnetic resonance imaging, positron emission tomography / computed tomography (PET / CT).

Treatment methods in childhood cancers are as follows; surgery, chemotherapy, radiotherapy and stem cell transplantation. Once diagnosed, oncologists and surgeons may choose one of these treatment options by mutual consultation or decide on a treatment method. Fractal analysis is a numerical as fractal dimension. Trabeculae are thin columns with numerous large spaces that give a honeycomb or spongy appearance of cancellous bone, which is also called trabecular bone or spongy bone. Previously, fractal analysis has been reported as a useful method to detect various diseases that affect the trabecular bone structure. Particularly in the field of dentistry, studies have shown that fractal analysis by the box-counting method can successfully evaluate trabecular changes in the mandible of patients with osteoporosis and periodontal diseases and in lactating women.

ELIGIBILITY:
Inclusion Criteria:

* to have been treated for any oncological diseases in childhood
* oncological treatment completed at least one year ago

Exclusion Criteria:

* ongoing oncological treatment
* patients who unwilling to participate to study

Ages: 6 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients received chemotherapy and radiotherapy for a Pediatric oncologic disease
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-08-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Bone Mineral Density (BMD) | Participants to undergo a single assessment; to be measured at least 1 year after completion of oncologic therapy
  Fractal Dimension of the mandibular bone in patients with pediatric oncologic diseases will be measured on dental panoramic images to asses bone mineral density of mandibula. Image J software will be used to Fractal Analysis measurements.

CONTACTS AND LOCATIONS:
Locations (1):
- Nuh Naci Yazgan University, Kayseri, Kocasinan, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
all types of data can be shared with other researchers.